CLINICAL TRIAL: NCT03057288
Title: Prospective Study Evaluating the Feasibility of Fiducial Markers Placement Under Echoendoscopy (EUS) Guidance for Patients With Esophageal or Rectal Cancer With an Indication of Radiotherapy
Brief Title: Prospective Study Evaluating the Feasibility of Fiducial Markers Placement for Patients With Esophageal or Rectal Cancer
Acronym: FIDECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société Française d'Endoscopie Digestive (Other)
Collaborators: Cook Group Incorporated (Industry)
Responsible Party: Principal Investigator, Chaput Ulriikka, Dr Ulriikka CHAPUT MD, Saint Antoine University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Etude SFED 115
Record Dates: First submitted 2017-02-09; First posted 2017-02-20 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Esophageal Neoplasm; Rectal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective study with one single group of 40 patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- fiducial markers placement (Experimental): Prospective study with one arm evaluating the feasibility of fiducial markers placement under echoendoscopic guidance, for patients with esophageal or rectal cancer
  Interventions: Device: fiducial markers placement

INTERVENTIONS:
Device: fiducial markers placement — The main objective of this study is to evaluate the feasibility of fiducial markers placement under EUS guidance for patients with esophageal or rectal cancer with an indication of radiotherapy

SUMMARY:
It is a multicenter prospective observational study including consecutive patients with esophageal tumor or rectum with indication for radiotherapy

The main objective of this study is to evaluate the feasibility of fiducial markers placement under EUS guidance. The evaluation criteria are:

* Success rate evaluation of the placement of two markers : one in the upper part of the tumor and one in the lower part. Success of the procedure will be evaluated by the endoscopist at the end of the procedure. Pictures of the markers will objectify the good placement of the markers.
* Complications (early within 24 hours and late complications) such as pain, bleeding, perforation, infection, migration of the markers
* The length of the procedure
* The costs (procedure, hospitalization)
* The clinical efficacy, by studying the decrease of the estimated target volume, the decrease of the dose delivered to the healthy tissue and the improvement of positioning of the irradiation beams by the radiotherapy technician
* The presence of the markers at the end of the radiotherapy

DETAILED DESCRIPTION:
* Rational Cancers of the rectum and esophagus affect 15 000 and 4300 people per year in France (TNCD, the national digestive cancer thesaurus). Their prognosis remains bleak, particularly due to late diagnosis, with a 5-year survival rate of 10% for cancers of the esophagus and 55% at 5 years for rectal cancers (TNCD). When diagnosed at an advanced stage (> T2 or N +), treatment with radiotherapy +/- chemotherapy is indicated. The precise definition of macroscopic tumor volume in radiotherapy represents an important difficulty because it is based on endoscopic and imaging data obtained under conditions different from those used in the preparation of radiotherapy treatment. A better definition of the target tumor volume using radiopaque markers known as fiducial markers would be likely to improve the efficacy and tolerance of this treatment, or even to allow additional irradiation that would be targeted more precisely on the tumor.
* Objectives :

The main objective of this study is to evaluate the feasibility of fiducial markers placement under EUS guidance.

The secondary objectives are to evaluate :

* Complications (early within 24 hours and late complications) such as pain, bleeding, perforation, infection, migration of the markers
* The length of the procedure
* The costs (procedure, hospitalization)
* The clinical efficacy, by studying the decrease of the estimated target volume, the decrease of the dose delivered to the healthy tissue and the improvement of positioning of the irradiation beams by the radiotherapy technician
* The presence of the markers at the end of the radiotherapy primary and secondary • Research methodology It is a prospective multicenter study, 18 centers will participate. Forty patients are to include over a period of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years
* Patients presenting an oesophageal or a rectal tumor passable with a linear echoendoscope
* TP> 60% et Platelets > 50 000/mm3
* No anticoagulant treatment or antiagregants being taken other than aspirin in the five days preceding the EUS
* Patient affiliated to a social security scheme (payee or beneficiary)
* Patient who signed a free and informed consent

Exclusion Criteria:

* Patient < 18 years
* Pregnant Woman
* Tumor stenosis impassable by the linear echoendoscope
* Patient participation refusal
* Patient under legal protection regime (guardianship / curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
Success rate evaluation of the placement of two fiducial markers | At the end of the endoscopic procedure, up to 2 hours
  One marker in the upper part of the tumor and one in the lower part. Success of the procedure will be evaluated by the endoscopist at the end of the procedure. Pictures of the markers will objectify the good placement of the markers.

SECONDARY OUTCOMES:
Complications (early within 24 hours and late complications) such as pain, bleeding, perforation, infection, migration of the markers | Day 1, Day 30 and Day 90
  phone contact clinical examination at Day 1, clinical examination at day 30 and at the end of the radiotherapy treatment (day 90)
The length of the procedure | the endoscopic procedure, up to120 minutes
  Duration in minutes of the endoscopic procedure
The costs (procedure, hospitalization) | up to two days of hospitalization without any complication
  sum of all costs : hospital stay, endoscopic procedure, fiducial markers
The clinical efficacy, by studying the decrease of the estimated target volume, the decrease of the dose delivered to the healthy tissue | Clinical examination with the radiotherapist, up to 30 minutes
  Before starting the radiotherapy, the target volume will be estimated with and without fiducial markers, thus estimating the decrease of the estimated target volume and the decrease of the dose delivered to the healthy tissue
The presence of the markers at the end of the radiotherapy | Clinical examination at the end of the radiotherapy with CT scan or MRI, up to 90 days
  Visualization of the fiducial markers on CT scan or MRI

CONTACTS AND LOCATIONS:
Overall Officials: Geoffroy VANBIERVLIET, M.D., Study Chair — Nice University hospital
Locations (1):
- Ulriikka CHAPUT, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Camus M, Karsenti D, Levy J, Moreno M, Coron E, Esch A, Williet N, Wangermez M, Koch S, Valats JC, Pioche M, Becq A, Vanbiervliet G, Audureau E, Huguet F, Chaput U. Success rate of fiducial marker placement for treatment of esophageal or rectal cancers: a prospective multicenter study (FIDECHO study) (with video). Gastrointest Endosc. 2025 Mar;101(3):570-577. doi: 10.1016/j.gie.2024.08.014. Epub 2024 Aug 20. PMID 39173781